CLINICAL TRIAL: NCT01789541
Title: Observational Prospective Case-control Study on Prevalence and Impact of Subclinical Hyperthyroidism in Patients Undergoing Atrial Fibrillation Ablation
Brief Title: Is a Low Thyreotropin Level Predictive of Recurrent Arrhythmia After Catheter Ablative Surgery?
Acronym: TABLAS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Giesecke, M.D, M.D., Karolinska Institutet
Other Study IDs: 3/9A
Record Dates: First submitted 2013-02-05; First posted 2013-02-12 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation; Subclinical Hyperthyroidism
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atrial fibrillation: Patients with atrial fibrillation undergoing ablation
- AV-nodal reentry tachycardia: Patients with AV-Nodal Reentry Tachycardia undergoing ablation

SUMMARY:
Overt hyperthyroidism (so-called "goiter" in lay language) is a hormonal disturbance that is known to increase the risk of atrial fibrillation (a common heart arrhythmia with potentially severe consequences) in some patients. Previous research has indicated that even slight elevations in thyroid hormone levels - so called subclinical hyperthyroidism - may increase this risk. When atrial fibrillation and overt hyperthyroidism are found simultaneously in a patient, the hormonal imbalance must be treated first in order to later resolve the arrhythmia. It is unclear whether this strategy holds true for subclinical hyperthyroidism. Our two hypotheses are: 1) Subclinical hyperthyroidism is more prevalent in patients admitted for atrial fibrillation ablation than in the population as a whole, and 2) Patients with subclinical hyperthyroidism and atrial fibrillation benefit less from ablation than others.

As a control group, we have chosen patients admitted for ablation of AV-nodal Reentry Tachycardia at the same clinics as the cases. No correlation has ever been shown between AV-nodal Reentry Tachycardia and hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation or AV-nodal reentry tachycardia
* Fulfills criteria for ablation (severe arrhythmia symptoms; for atrial fibrillation patients, having tried at least one antiarrhythmic agent with poor effect)
* Admitted for ablation for the first time
* Has left blood samples for thyroid status (TSH, free T4, free T3)

Exclusion Criteria:

* Atrial flutter
* Overt hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation (cases) or AV-nodal reentry tachycardia (controls)
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of subclinical hyperthyroidism in patients undergoing atrial fibrillation ablation | 1 day (Measured upon inclusion)

SECONDARY OUTCOMES:
Recurrent atrial fibrillation after ablation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Rosenqvist, Professor, Study Chair — Karolinska Institutet, Institutionen för kliniska vetenskaper vid Danderyds sjukhus
Locations (2):
- Sweden (2):
  - Stockholm Arrhythmia Center, Stockholm
  - Hjärtkliniken, Karolinska Universitetssjukhuset Huddinge, Stockholm